CLINICAL TRIAL: NCT02333032
Title: Evaluation of Biomechanical and Functional Effects of a Positive Slope Treadmill Training in Individuals After Stroke.
Brief Title: Effects of a Positive Slope Treadmill Training in Individuals After Stroke. (Hemislope)
Acronym: Hemislope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01500-47
Record Dates: First submitted 2014-12-24; First posted 2015-01-07 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: randomised controlled study experimental group : training with slope N=15 control group training with no slope N=15
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemiplegic patient (Experimental)
  Interventions: Other: Inclined treadmill training

INTERVENTIONS:
Other: Inclined treadmill training

SUMMARY:
The main objective of this study is to determine if a single session of treadmill training with a positive slope improves the kinematic parameters of the hip, knee and ankle on the paretic lower limb.

Secondarily we will quantify the efficiency of a such training on kinetic and functional parameters.

DETAILED DESCRIPTION:
comparison between patients having a single session of treadmill training with slope and those having a single session of treadmill training with no slope

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patient
* capacity to walk during 20 minutes without technical assistance

Exclusion Criteria:

* patient with bilateral brain lesions
* previous orthopedic surgery
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
kinematic gait parameters | One year
  angles quantification of lower limbs joints
cinetic gait parameters | one year
  moments and joints power quantification in the lower limb

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France

IPD SHARING:
Plan to Share IPD: No